CLINICAL TRIAL: NCT02075762
Title: Comparison of Transbronchial, Cryoprobe, and VATS Biopsy for the Diagnosis of Interstitial Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00083791
Record Dates: First submitted 2013-09-03; First posted 2014-03-03 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Transbronchial biopsy (Active Comparator): S-TBBx will be performed using standard biopsy forceps (Boston Scientific, Natick, MA) - 2.0mm diameter.
  Interventions: Procedure: Transbronchial biopsy
- Cryoprobe biopsy (Active Comparator): C-TBBx will be performed using the cryoprobe (ERBE, Tubingen, Germany) -1.9 mm diameter, 78cm in length. This cryoprobe is routinely used in the bronchoscopy suite for carcinoma-TBBX; therefore it is a technique already employed by the interventional pulmonologists who are familiar with its use.
  Interventions: Procedure: Cryoprobe biopsy
- VATS biopsy (Active Comparator): Once the biopsies are obtained by the interventional pulmonologist, the thoracic surgeon will perform VATS biopsy. Following their procedure, subjects will be monitored in the post-anesthesia care unit as per standard of care. As part of their ongoing follow-up care, all subjects will be monitored for any adverse events that may have resulted from either the surgical or bronchoscopic procedure, specifically bleeding or pneumothorax.
  Interventions: Procedure: VATS biopsy

INTERVENTIONS:
Procedure: Transbronchial biopsy
  Arms: Transbronchial biopsy
Procedure: Cryoprobe biopsy
  Arms: Cryoprobe biopsy
Procedure: VATS biopsy
  Arms: VATS biopsy

SUMMARY:
The objective of this study is to compare the sample size, architectural preservation and diagnostic yield of bronchoscopic cryo-probe transbronchial lung biopsy (C-TBBx) in comparison to bronchoscopic standard transbronchial lung biopsy (S-TBBx) and Video-Assisted Thoracoscopic Surgery (VATS) lung biopsy for the diagnosis of interstitial lung disease (ILD).

DETAILED DESCRIPTION:
This is a prospective cohort study in which 20 subjects that have suspected ILD who are undergoing non-emergent surgical biopsy will be enrolled.

Patients who have been referred to the thoracic surgery service for VATS biopsy to diagnose suspected ILD and meet basic inclusion/exclusion criteria will be approached by the study investigators and informed of the study. An informed consent will be obtained during the clinic visit with the thoracic surgeon.

At the beginning of the surgical procedure, under general anesthesia in the operating room, patients will undergo flexible bronchoscopy through the endotracheal tube and obtain 10 standard transbronchial biopsies (S-TBBx) and 5 Cryoprobe biopsies (C-TBBx) with fluoroscopic guidance. S-TBBx will be performed using standard biopsy forceps (Boston Scientific, Natick, MA) - 2.0mm diameter. C-TBBx will be performed using the cryoprobe (ERBE, Tubingen, Germany) -1.9 mm diameter, 78cm in length. This cryoprobe is routinely used in the bronchoscopy suite for other applications such as foreign body removal and local treatment of carcinoma; therefore it is a technique already employed by the interventional pulmonologists who are familiar with its use. Once the biopsies are obtained by the interventional pulmonologist, the thoracic surgeon will perform video-assisted thoracoscopic biopsy (VATS) biopsy. Following their procedure, subjects will be monitored in the post-anesthesia care unit as per standard of care. As part of their ongoing follow-up care, all subjects will be monitored for any adverse events that may have resulted from either the surgical or bronchoscopic procedure, specifically bleeding or pneumothorax.

All biopsy samples will be analyzed by a specialist in pulmonary pathology.

The number and size of all biopsies, architectural preservation of the airways/alveoli, and pathological diagnosis will be reported by the pathologist. Diagnostic yield will be calculated for each biopsy technique and compared

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Scheduled VATS biopsy for suspected ILD as part of standard medical care
* Negative pregnancy test
* Mentally capable of understanding study procedures

Exclusion Criteria:

* A disease or condition that interferes with safe completion of the study including:

  * Platelet count < 50,000 Coagulopathy defined as an International
  * Normalized Ratio (INR) > 1.5, or discontinuation of ticagrelor or clopidogrel within 5 days of procedure.
  * Hemodynamic instability with systolic blood pressure <90 mmHg or heart rate > 120 beats/min, unless deemed to be stable with these values by the surgical or interventional pulmonary attending physicians
  * Hypoxemia with pulse oximetry values <88% or partial pressure of oxygen in arterial blood (PaO2) < 60 on baseline oxygen requirements
* Concurrent participation in another study involving investigational drugs or investigational medical devices

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Comparison of biopsy technique | Data will be measured one week post procedure
  The number and size of all biopsies, architectural preservation of the airways/alveoli, and pathological diagnosis will be reported by the pathologist. Diagnostic yield will be calculated for each biopsy technique and compared

CONTACTS AND LOCATIONS:
Overall Officials: Lonny Yarmus, Principal Investigator — Johns Hopkins SOM
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States